CLINICAL TRIAL: NCT05242419
Title: A Multi-center, Randomized, Double-blinded, Placebo-controlled Study of Huperzine A Injection in Reducing Postoperative Delirium in Elderly Patients Undergoing Non-cardiac Surgery
Brief Title: A Study of Huperzine A Injection in Reducing Postoperative Delirium in Elderly Patients Undergoing Non-cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Affiliated Wenling Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Ting Li, Principal Investigator, Second Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SSJJZ-WW-01
Record Dates: First submitted 2022-01-09; First posted 2022-02-16 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Injection; Non-cardiac Surgery; Delirium in Old Age; Post Operative Delirium
Keywords: Huperzine A Injection; postoperative delirium; Non-cardiac Surgery; Elderly Patients
MeSH Terms: conditions — Emergence Delirium | interventions — Sodium Chloride; huperzine A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Huperzine A Injection
  Interventions: Drug: Huperzine A Injection
- Control group (Placebo Comparator): 0.9% Sodium Chloride Injection
  Interventions: Drug: Sodium Chloride Injection

INTERVENTIONS:
Drug: Sodium Chloride Injection — 0.9% Sodium Chloride Injection
  Arms: Control group
Drug: Huperzine A Injection — Huperzine A Injection
  Arms: Treatment group

SUMMARY:
To observe and study the clinical effect of Huperzine A Injection on reducing postoperative delirium in elderly patients undergoing non-cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

* ≥ 75 years old.
* Comply with the indication of non-cardiac surgery under general anesthesia.
* Anesthesia grade of American Society of Anesthesiologist (ASA) as III~IV grade.
* The estimated operation time ≥ 2 hours.
* Voluntarily sign the informed consent form.

Exclusion Criteria:

* Patients with impaired renal function (Cr is 1.5 times higher than the upper limit of the normal value of the central laboratory) or abnormal liver function (Alanine aminotransferase(ALT) and Aspartate aminotransferase(AST) are 2 times higher than the upper limit of the normal value of the central laboratory).
* Patients who are positive for infectious diseases.
* Patients accompanied with central nervous system injury.
* Patients with previous history of delirium and epilepsy, long-term use of psychoactive drugs or preoperative assessment of delirium.
* Patients who involved diseases with drug taboos, bronchial asthma, mechanical intestinal obstruction and urinary tract obstruction, or serious systemic diseases, especially circulatory diseases: such as myocardial infarction, heart failure, angina pectoris, history of sinus bradycardia.
* Patients who are known to be allergic to narcotic drugs or Huperzine A Injection, or must use drugs that are not compatible with Huperzine An Injection.
* patients who participated in other clinical trials within 3 months before this study, for any reason, who could not tolerate the test or cooperate with the examination, or who has any aphasia, audio-visual dysfunction, etc.
* the investigators think that the patients is not suitable to participate in this study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium within 7 days after operation | 7 days after operation
  Delirium will be evaluated by The 3-dimensional Confusion Assessment Method(3D-CAM) and delirium rating scale-revised-98(DRS-R-98) scale form.

SECONDARY OUTCOMES:
type of delirium | evaluated at screening, 24 hours, 48 hours, 72 hours after operation
  diagnosed by delirium rating scale-revised-98(DRS-R-98) scale form
severity of delirium | evaluated at screening, 24 hours, 48 hours, 72 hours after operation
  diagnosed by delirium rating scale-revised-98(DRS-R-98) scale form
duration of delirium | evaluated at screening, 24 hours, 48 hours, 72 hours after operation
  diagnosed by delirium rating scale-revised-98(DRS-R-98) scale form
length of hospital stay | from the day of operation to the day of discharge, around 7 to 14 days
  total number of days of hospital stay
Economic indicators (total hospitalization cost, anesthesia cost, operation cost). | through study completion, up to 2 months
  costs at hospital
Occurrence of complications | through study completion, up to 2 months
  pulmonary infection, myocardial infarction, renal failure, gastrointestinal bleeding, etc.
Incidence of Mortality | the day of hospital discharge, and the day of follow-up, around 30 days after discharge
  rate of Mortality during the hospital stay and follow-up within 30 days after discharge
the total score of Mini-mental State Examination scale | evaluated at screening, 72 hours after operation, and the day of follow-up, around 30 days after discharge
  Mini-mental State Examination scale
the score of EuroQol (EQ-5D) scale | 96 hours after operation, the day of hospital discharge, and the day of follow-up, around 30 days after discharge
  EQ-5D scale

CONTACTS AND LOCATIONS:
Overall Officials: Ting Li, MD. PhD, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The 2nd Second Affiliated Hospital of WMU Phase I Clinical Trial Unit /Center Of Bioequivalence Study, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No